CLINICAL TRIAL: NCT04320446
Title: Caffeine Increases Maximal Fat Oxidation During Exercise in Endurance-trained Men: is There a Diurnal Variation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Jonatan Ruiz Ruiz, Associate professor, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: Nº 507/CEIH/2018
Record Dates: First submitted 2020-03-19; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Energy Metabolism; Athletic Performance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeine (Experimental): A dose of 3 mg/kg of caffeine (i.e. a vegetable extraction from green coffee beans, Harrison Sport Nutrition®, Spain) was ingested before the beginning of each test.
  Interventions: Behavioral: Test in the morning; Behavioral: Test in the afternoon
- Placebo (Placebo Comparator): A dose of 3 mg/kg of placebo (i.e. 100% purity microcrystalline cellulose, Acofarma, Spain) was ingested before the beginning of each test.
  Interventions: Behavioral: Test in the morning; Behavioral: Test in the afternoon

INTERVENTIONS:
Behavioral: Test in the morning — The exercise test was performed between 8 a.m and 11 a.m
  Other Names: MFO-morning, Fatmax-morning, and VO2max-morning
Behavioral: Test in the afternoon — The exercise test was performed between 5 p.m. and 8 p.m.a
  Other Names: (MFO-afternoon, Fatmax-afternoon, and VO2max-afternoon

SUMMARY:
Maximal fat oxidation during exercise (MFO) and the intensity of exercise that elicits MFO (Fatmax) has been recognized as potential determinants of endurance performance.

The purpose of this study was to determine the possible interaction between the effects of diurnal variation (morning vs. afternoon) and caffeine ingestion on MFO, Fatmax and VO2 max in endurance-trained men. Specifically, the investigators sought to elucidate whether the stimulant actions of caffeine could reverse the decrements of MFO and Fatmax observed in the morning.

DETAILED DESCRIPTION:
Body weight, height, body composition (DXA), exercise test (MFO and VO2max assessment) will be measured during the 4 evaluations.

Participants were randomized into 4 exercise test conditions:

1. Exercise test in the morning with placebo intake
2. Exercise test in the evening with placebo intake
3. Exercise test in the morning with caffeine intake
4. Execrise test in the evening with caffeine intake

ELIGIBILITY:
Inclusion Criteria:

* Having a body mass index (BMI) ranged from 18.5 to 28 kg/m2
* not suffering any specific disease which can be aggravated by physical exercise
* having previous experience in endurance training (i.e. self-reporting at least 2 years of cycling or running training including more than 3 training sessions/week).
* Participant must be capable and willing to provide consent, understand exclusion criteria, instructions and protocols.

Exclusion Criteria:

* Being smoker
* Taking medication or drugs
* Any non-controlled medical condition which could influence results or could be worsened by the participation in the study
* Are deemed unsuitable by the investigator for any other reason, that prevent data collection.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
MFO | Through study completion, an average of 1 month
  Maximal fat oxidation during exercise

SECONDARY OUTCOMES:
FATmax | Through study completion, an average of 1 month
  The intensity of exercise that elicits MFO
VO2max | Through study completion, an average of 1 month
  Cardiorrespiratory fitness measured by maximal oxygen uptake

CONTACTS AND LOCATIONS:
Overall Officials: Jonatan Ruiz Ruiz, Dr., Principal Investigator — Universidad de Granada
Locations (1):
- Instituto Mixto Universitario Deporte Salud, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez-Maldonado M, Jurado-Fasoli L, Del Coso J, R Ruiz J, Amaro-Gahete FJ. Caffeine increases maximal fat oxidation during a graded exercise test: is there a diurnal variation? J Int Soc Sports Nutr. 2021 Jan 7;18(1):5. doi: 10.1186/s12970-020-00400-6. PMID 33413459